CLINICAL TRIAL: NCT02677636
Title: A Phase 3, Double-Blind, Randomized, Vehicle-Controlled, Multicenter, Parallel Group Evaluation of the Efficacy and Safety of MSRD-100 in Subjects >=3 Months of Age With Atopic Dermatitis
Brief Title: Efficacy and Safety Study of MSRD-100 in Subjects With Atopic Dermatitis >=3 Months of Age and Older
Acronym: MSRD-100
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M169981002
Record Dates: First submitted 2016-01-27; First posted 2016-02-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Atopic Dermatitis
Keywords: Dermatitis, Atopic; Eczema; Dermatitis; Pruritus; Genetic Diseases, Inborn; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases; Skin Diseases, Eczematous; Skin Diseases, Genetic; Skin Diseases; Itching; Rash; Steroid
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Pruritus; Genetic Diseases, Inborn; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases; Skin Diseases, Eczematous; Skin Diseases, Genetic; Skin Diseases; Exanthema | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSRD-100 (Experimental): MSRD-100 is a topical gel with an active ingredient in a vehicle. Excipients are purified water, propylene glycol, polysorbate 20, benzyl alcohol, edetate disodium, diethylene glycol monoethyl ether and hydroxyethyl cellulose. Application is twice daily for 28 days.
  Interventions: Drug: MSRD-100
- Placebo Comparator (Placebo Comparator): The vehicle is a topical gel and contains excipients of the formulation: purified water, propylene glycol, polysorbate 20, benzyl alcohol, edetate disodium, diethylene glycol monoethyl ether and hydroxyethyl cellulose. It does not contain the active ingredient MSRD-100. Application is twice daily for 28 days.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: MSRD-100 — MSRD-100 is a topical gel.
  Other Names: Active
  Arms: MSRD-100
Drug: Vehicle — Vehicle is a topical gel without the active ingredients in MSRD-100
  Other Names: Placebo
  Arms: Placebo Comparator

SUMMARY:
This is a double-blind, randomized, vehicle-controlled, multi-center, parallel group Phase 3 study of MSRD-100 in the treatment of atopic dermatitis in subjects aged 3 months and up

DETAILED DESCRIPTION:
This is a 4-week efficacy, safety and tolerability study of MSRD-100 applied twice daily for 4 weeks compared to its vehicle among subjects ≥3 months of age in the treatment of atopic dermatitis covering ≥5% body surface area.

The study will consist of up to 4 visits which includes Screening - Visit 1 (Screening), Baseline - Visit 2 , Visit 3 (Day 14), and an End of Treatment/Final Study Visit - Visit 4 (Day 28).

Study IDs M169981001 and M169981002 are two identical studies being run in parallel with different study sites.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects who are male or female, ≥3 months of age on the date of Baseline Visit.
2. Subjects with a diagnosis of atopic dermatitis, active inflammation and meeting the Hanifin and Rajka Diagnosis Criteria for atopic dermatitis.
3. Subjects must have an Investigator Global Assessment (IGA) score of ≥2 at baseline.
4. Subjects who have atopic dermatitis covering ≥5% Body Surface Area (BSA) excluding the eyelids, perioral area, around the nostrils, and in the diaper area (for subjects who wear diapers or plastic pants).
5. Subjects who have atopic dermatitis with a sign and symptom score ≥ 2 on the following three signs and symptoms: erythema, infiltration/papulation, and erosion/oozing/crusting present in at least one body surface area affected.

Key Exclusion Criteria:

1. Unstable course of atopic dermatitis (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to baseline.
2. Concurrent conditions and history of other diseases.
3. Used any of the following treatments within the indicated washout period before the baseline visit or those who would require the following during the study.
4. Subjects who require treatment with any other topical or systemic therapy for the study disease other than bland emollients in untreated areas of disease.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of subjects with treatment success in the MSRD-100 and vehicle group | Visit 4 (Day 28)
  Treatment success is defined as an Investigator Global Assessment (IGA) score of clear or almost clear and a minimum of a 2-grade improvement in IGA score from baseline plus no worsening on any of the signs present at baseline.
  The primary endpoint is a composite of: (1) the IGA score of clear or almost clear as well as subjects having a minimum two point improvement on the IGA, plus (2) no worsening of any of the signs present at baseline.

SECONDARY OUTCOMES:
Compare the proportion of subjects with an IGA score of 0 or 1 between the MSRD-100 and vehicle at Visit 4 | Visit 4 (Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuligowski, MD, PhD, MBA, Study Director — Study Director